CLINICAL TRIAL: NCT00750685
Title: Study of the Safety and Effectiveness of the Mentor Becker Expander/Breast Implant in Subjects Who Are Undergoing Primary Breast Reconstruction
Brief Title: Study of the Mentor Becker Expander/Breast Implant in Subjects Who Are Undergoing Primary Breast Reconstruction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Terminated
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-101-0501-8; Becker Study
Expanded Access: NCT01000012 (No longer available)
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Breast Reconstruction
Keywords: Primary Breast Reconstruction
MeSH Terms: interventions — Breast Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reconstruction (Other): The study population will consist of women aged 18 or over who are undergoing primary breast reconstruction.
  The Reconstruction cohort will include subjects with loss of breast tissue due to mastectomy, contralateral breast for post-reconstruction symmetry or subjects with deformities secondary to disease, malignancy, trauma, and congenital deformity. Subjects in this cohort cannot have been implanted with breast implants, but may have tissue expanders. A Becker implant is considered a tissue expander until the port and fill tube have been removed. Women who undergo surgery primarily for a mastopexy will not be part of the reconstruction cohort.
  Interventions: Device: Mentor Smooth Becker 50 Expander/Breast Implant

INTERVENTIONS:
Device: Mentor Smooth Becker 50 Expander/Breast Implant — The Mentor Becker Expander/Breast Implant is comprised of two components: the Becker implant and the injection dome/fill tube. The breast implant is available in a smooth surface. It has a low bleed, gel-filled outer lumen and an adjustable saline-fillable inner lumen. The silicone elastomer fill tube is pre-inserted into the dual self-sealing valve system at the time of manufacture and is joined to the injection dome by the connector system at the time of surgery. The inner lumen can be gradually filled with saline over an extended period of time via the fill tube by injecting saline through the injection dome. Once expanded to the desired volume, the fill tube and injection dome are removed through a small incision under local anesthetic, and the prosthesis remains in position as a breast implant.
  Other Names: Breast Implant; Double-Lumen Breast Implant; Becker Implant

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the Becker Expander/Breast Implant in women who are undergoing primary breast reconstruction. Safety information on the rate of complications, such as infection will be collected, and used to help determine device safety. These implants are investigational devices.

Approximately 300 patients at centers across the United States will be enrolled in this research study, by up to 30 sites. These patients will be implanted with Becker Expander/Breast Implant and monitored for 10 years to collect information on risks associated with the implant surgery as well as changes in the way these patients feel about themselves.

DETAILED DESCRIPTION:
Silicone gel-filled breast implants were introduced in the early sixties and were in wide-scale distribution by the time the Medical Device Amendments to the Food Drug and Cosmetic Act was passed in 1976. In 1983, gel-filled breast implants were designated as Class III devices requiring premarket approval. In May 1990, the Food and Drug Administration (FDA) published a proposed request (515(b)) for Pre-market Approval Applications (PMA) and in April 1991 published the final request. This final publication put manufacturers of gel-filled breast implants on notice that for continued marketing of gel-filled breast implants, a PMA was due to FDA in 90 days from the final publication date.

A pre-market approval (PMA) for the Mentor gel-filled breast implants was filed with the FDA in July 1991. At the FDA General and Plastic Surgery Advisory Committee meeting in November 1991, the committee recommended the submission of additional information to establish the safety and effectiveness of gel-filled breast implants.

In January 1992, the FDA Commissioner announced a voluntary moratorium of the sale of gel-filled breast implants to allow the advisory panel time to assess additional information. In April 1992, the moratorium was lifted but only for reconstruction and revision subjects. Every subject implanted had to be part of an adjunct study, in addition to being offered participation in a registry of gel-filled breast implant subjects. In order to be implanted with gel-filled implants for augmentation, women had to be enrolled in an IDE clinical trial.

A PMA for Mentor's MemoryGel™ Silicone Gel-Filled breast implants (which did not include the Becker Expander/Breast Implants) was subsequently filed with FDA in December 2003, and approved in November 2006 (P030053). As a condition of approval of P030053, new enrollment in Mentor's Adjunct Study has ceased, and women no longer have access to the Becker Expander/Breast Implants.

This study is designed to evaluate the safety and effectiveness of Mentor's Becker Expander/Breast Implants for primary breast reconstruction

ELIGIBILITY:
Inclusion Criteria:

Patients will be allowed to enter the study if the following inclusion criteria are met:

* Subject is genetic female, 18 years of age or older
* A candidate for primary breast reconstruction for cancer, trauma, surgical loss of breast tissue due to mastectomy, malignancy, contralateral post-reconstruction symmetry, or congenital deformity, including asymmetry
* Signs the Informed Consent
* Agrees to return device to Mentor if explant necessary
* Agrees to comply with follow-up procedures, including returning for all follow-up visits

Exclusion Criteria:

Patients will not be allowed to enter the study if they have any of the following exclusion criteria:

* Subject is pregnant
* Has nursed a child within three months of study enrollment
* Been implanted with any silicone implant other than breast implants (e.g. silicone artificial joints or facial implants)
* Confirmed diagnosis of the following rheumatic diseases or syndromes: SLE, Sjogren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondylarthropathies, any other inflammatory arthritis, fibromyalgia, or chronic fatigue syndrome
* Currently has a condition that could compromise or complicate wound healing (except reconstruction subjects)
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics which are clinically incompatible with implant (e.g. tissue damage resulting from radiation, inadequate tissue, or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physicians(s), may constitute an unwarranted surgical risk
* Anatomic or physiologic abnormality which could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Premalignant breast disease without a subcutaneous mastectomy
* Untreated or inappropriately treated breast malignancy, without mastectomy
* Are HIV positive
* Work for Mentor or the study doctor or are directly-related to anyone that works for Mentor or the study doctor
* Implanted metal or metal devices, history of claustrophobia or other condition that would make a MRI scan prohibitive
* Surgeon intending to use the device for tissue expansion only

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2014-03-04 (Actual); Study Completion 2014-03-04 (Actual)

PRIMARY OUTCOMES:
Safety will be determined by the incidence, severity, method of resolution, and duration for all adverse events on a per implant and per subject basis. | 10 years
Effectiveness will be determined by changes in chest circumference and bra and cup size. | 10 years

SECONDARY OUTCOMES:
Effectiveness will also be determined by changes in validated Quality of Life instrument ratios. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Janet Vargo, Study Director — Mentor Worldwide, LLC